CLINICAL TRIAL: NCT00744172
Title: Finhyst 2006: Incidence, Methods, Complications and Effect on Quality of Life of Hysterectomies in Finland in 2006
Brief Title: Finhyst 2006: Study on Morbidity of Hysterectomies in Finland
Acronym: Finhyst 2006
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Society for Gynecological Surgery in Finland (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Paivi Harkki, MD PhD, Society for Gynecological Surgery in Finland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Finhyst 2006
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Morbidity of Hysterectomy
Keywords: hysterectomy; vaginal; laparoscopy; abdominal; complication; quality of life; cost-effectiveness; Morbidity of three types of hysterectomy
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- I (Active Comparator): laparoscopy
  Interventions: Procedure: laparoscopy
- 2 (Active Comparator): vaginal
  Interventions: Procedure: vaginal
- 3 (Active Comparator): abdominal
  Interventions: Procedure: abdominal

INTERVENTIONS:
Procedure: laparoscopy — laparoscopic hysterectomy
  Arms: I
Procedure: vaginal — vaginal hysterectomy
  Arms: 2
Procedure: abdominal — abdominal hysterectomy
  Arms: 3

SUMMARY:
The purpose of this study is to analyze prospectively all hysterectomies performed in Finland for benign indications including all 46 public hospitals performing hysterectomies and also 7 private clinics. Hypothesis is that vaginal and laparoscopic hysterectomies are safe and cost-effective methods of hysterectomy.

DETAILED DESCRIPTION:
This Finhyst 2006 study evaluates nationwidely methods, indications, concomitant procedures, complications, hospital stay and convalescence time of all types of hysterectomies with questionnaires filled by doctors and patients. In addition, in the area of Helsinki University Central Hospital also the effect of quality of life and cost-effectiveness is studied.

ELIGIBILITY:
Inclusion Criteria:

* Bening indications for hysterectomy

Exclusion Criteria:

* Malignant indications for hysterectomy
* Postpartum hysterectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5279 (Actual)
Dates: Start 2006-01; Primary Completion 2006-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety of hysterectomy | 1.1-31.12.2006

SECONDARY OUTCOMES:
Cost-effectiveness | 1.1.-31.12.2006

CONTACTS AND LOCATIONS:
Overall Officials: Päivi SM Härkki, MD, Study Director — Member of Society of Gynecological Surgery in Finland
Locations (1):
- Helsinki University Central Hospital, Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Makinen J, Brummer T, Jalkanen J, Heikkinen AM, Fraser J, Tomas E, Harkki P, Sjoberg J. Ten years of progress--improved hysterectomy outcomes in Finland 1996-2006: a longitudinal observation study. BMJ Open. 2013 Oct 28;3(10):e003169. doi: 10.1136/bmjopen-2013-003169. PMID 24165027
- [Derived] Brummer TH, Heikkinen AM, Jalkanen J, Fraser J, Makinen J, Tomas E, Seppala T, Sjoberg J, Harkki P. Antibiotic prophylaxis for hysterectomy, a prospective cohort study: cefuroxime, metronidazole, or both? BJOG. 2013 Sep;120(10):1269-76. doi: 10.1111/1471-0528.12178. Epub 2013 Jun 21. PMID 23786166
- [Derived] Brummer TH, Heikkinen A, Jalkanen J, Fraser J, Makinen J, Tomas E, Seppala T, Sjoberg J, Harkki P. Pharmaceutical thrombosis prophylaxis, bleeding complications and thromboembolism in a national cohort of hysterectomy for benign disease. Hum Reprod. 2012 Jun;27(6):1628-36. doi: 10.1093/humrep/des103. Epub 2012 Mar 14. PMID 22422792